CLINICAL TRIAL: NCT02203188
Title: Effect of Debridement-scaling on the Relief of Dry Eye Signs and Symptoms in Sjogren's Syndrome
Acronym: TOYOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Sjogren's Society of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20000
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lid debridgement scaling (Experimental): Perform lid debridgement scaling
  Interventions: Procedure: Lid debridgement scaling
- Control (No Intervention): No Treatment

INTERVENTIONS:
Procedure: Lid debridgement scaling
  Arms: Lid debridgement scaling

SUMMARY:
Sjogren's Syndrome is an autoimmune condition in which the body attacks its own glands in the body. Some of these glands are responsible for providing lubrication for the eye. As a result, individuals with Sjogren's Syndrome often experience dry eye. Recently, a study had shown that dry eye symptoms were improved by removing debris and old skin cells along the eyelid margin. This technique is called eyelid debridement-scaling. The purpose of this study is to determine how well this technique works in improving dry eye signs and symptoms in individuals with Sjogren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is diagnosed with Sjogren's Syndrome;
* Meibomian gland score of ≤ 9 (out of 15);
* OSDI ≥ 23;
* Willing to maintain the use of OTC medications throughout the course of the study
* Have not worn contact lenses within the past 3 years

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active* ocular disease and/or infection;
* Has a systemic condition, other than Sjogren's Syndrome and its associated conditions, that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications, other than those indicated for Sjogren's Syndrome and its associated conditions, that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment;
* Is aphakic;
* Has undergone refractive error surgery; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Meibomian gland score (MGS) | Baseline
  Prior to treatment (if applicable). Scale 0-3. 0: no secretion, 1: inspissated (toothpaste), 2: cloudy with debris, 3: clear
Meibomian gland score (MGS) | 1 month after baseline and/or treatment
  Scale 0-3. 0: no secretion, 1: inspissated (toothpaste), 2: cloudy with debris, 3: clear
SICCA Ocular Staining Score | Baseline
  Prior to treatment (if applicable). Based on corneal and conjunctival staining. Total scores range 0 to 12 with 0 being no staining and 12 being high staining.
SICCA Ocular Staining Score | 1 month after baseline and/or treatment
  Based on corneal and conjunctival staining. Total scores range 0 to 12 with 0 being no staining and 12 being high staining.
Ocular Surface Disease Index Score (OSDI) | Baseline
  Prior to treatment (if applicable). The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 to 100.
Ocular Surface Disease Index Score (OSDI) | 1 month after baseline/treatment
  The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 to 100.
Meibomian gland yielding liquid secretions (MGYLS) | Baseline
  Prior to treatment (if applicable). MGYLS is the number of glands with MGS grade 2 or higher.
Meibomian gland yielding liquid secretions (MGYLS) | 1 month after baseline/treatment
  MGYLS is the number of glands with MGS grade 2 or higher.
Symptom Assessment iN Dry Eye score | Baseline
  Prior to treatment (if applicable). A short questionnaire based on a visual analog scale (VAS) to quantify the frequency and severity of symptoms of dry eye syndrome. The "Symptom Assessment iN Dry Eye" (SANDE) questionnaire utilizes a 100 mm horizontal VAS technique to quantify patient symptoms of ocular dryness and/or irritation.
Symptom Assessment iN Dry Eye score | 1 month after baseline and/or treatment
  A short questionnaire based on a visual analog scale (VAS) to quantify the frequency and severity of symptoms of dry eye syndrome. The "Symptom Assessment iN Dry Eye" (SANDE) questionnaire utilizes a 100 mm horizontal VAS technique to quantify patient symptoms of ocular dryness and/or irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — CCLR, University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada